CLINICAL TRIAL: NCT07256366
Title: How Reliable Are Routine Radiological Imaging Methods in Diagnosing Lumbosacral Transitional Vertebrae and Identifying the Pathological Disc Level?
Status: Not yet recruiting | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Other Study IDs: MarmaraU-FTR-OK-2
Record Dates: First submitted 2025-11-20; First posted 2025-12-01 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Lumbosacral Transitional Vertebrae; Thoracolumbar Transitional Vertebra; Vertebral Level Misidentification; Lumbar Radiculopathy; Spinal Imaging Accuracy
Keywords: LSTV; TLTV; lomber rib; spinal imaging accuracy; transitional vertebrae; vertebral level misidentification
MeSH Terms: conditions — Radiculopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- GROUP 1: Patients who applied to the outpatient clinic with complaints of back and leg pain

SUMMARY:
The aim of this study is to evaluate how accurately transitional vertebrae can be identified using routinely employed clinical imaging methods, including thoracolumbar direct radiography and lumbar MRI with axial and sagittal sequences. The study also seeks to determine how anatomical markers commonly used in the literature for vertebral level identification correspond to vertebral levels in the Turkish population, and whether a new potential relationship between these anatomical markers can be identified to improve accurate vertebral numbering. Additionally, the study will assess the relationship between thoracolumbar transitional vertebra (TLTV) and lumbosacral transitional vertebra (LSTV) variations, and ultimately aims to provide new data to determine which imaging-based approach offers the highest diagnostic accuracy.

DETAILED DESCRIPTION:
Lumbosacral transitional vertebrae (LSTV) include morphological variants in which L5 is partially or completely fused with the sacrum (sacralization), or in which S1 assumes additional lumbar characteristics (lumbarization). The most commonly used classification is the Castellvi system, which categorizes these variations from Type I to Type IV. Based on data from the past decade, the prevalence of LSTV ranges between 7% and 36%. LSTV may restrict motion at the transitional segment and consequently lead to disc degeneration in adjacent levels. One study reported that the Pfirrmann grade of the disc above the transitional vertebra was significantly higher in individuals with LSTV. The most reliable method for diagnosing LSTV is counting vertebrae caudally from the C2 vertebra on whole-spine imaging. Since the presence of LSTV can result in incorrect vertebral level identification during surgical or interventional procedures, recognizing these variations is essential.

Transitional segments located in the thoracolumbar junction that display both thoracic and lumbar characteristics are defined as thoracolumbar transitional vertebrae (TLTV). TLTV commonly involves atypical rib formation at the last thoracic or first lumbar vertebrae. The presence of a 13th rib-also termed a lumbar rib-is another variant that complicates vertebral level identification. In radiography, the last vertebra with a true rib is generally accepted as T12, and lumbar vertebrae are counted accordingly. However, in some individuals, the transverse process of the first lumbar vertebra develops a rib-like morphology. This structure is referred to as a lumbar rib and may create ambiguity during lumbar level identification on radiographs. Although numerous studies have examined the prevalence and clinical implications of LSTV, data on TLTV remain insufficient.

Various imaging modalities and anatomical markers have been used for detecting transitional vertebrae. The most reliable method for identifying both LSTV and TLTV is whole-spine MRI or CT imaging that allows vertebral counting from C2 caudally. This approach directly reveals segmental anomalies and numbering variations. Although anatomical markers such as the aortic bifurcation, inferior vena cava bifurcation, right renal artery, and conus medullaris have been proposed for determining lumbar vertebral levels, their anatomical variability limits their reliability, particularly when used in isolation. Moreover, studies have shown that the position of these markers shifts depending on the presence of transitional vertebrae: markers tend to be positioned more caudally in sacralized vertebrae and more cranially in lumbarized vertebrae.

In this cross-sectional study, patients presenting with low back and leg pain to the Algology Division of the Department of Physical Medicine and Rehabilitation at Marmara University, who are diagnosed with lumbar radicular pain based on clinical evaluation and MRI, will be assessed. Demographic data, including age, sex, height, weight, and body mass index, will be recorded.

In the first stage of evaluation, the level of the disc herniation responsible for lumbar radicular pain will be determined on routine lumbar MRI sequences using anatomical markers described in the literature (right renal artery, conus medullaris, aortic and inferior vena cava bifurcations). Thoracolumbar and lumbosacral two-view radiographs will also be evaluated to identify transitional vertebrae and to note the presence of lumbar ribs, rudimentary thoracic ribs, or other costal anomalies. For each anatomical marker, the disc level suggested by that marker will be recorded separately, and the level indicated by the majority of markers will also be noted. If a transitional vertebra is identified on radiographs, the disc level determined on MRI will be revised accordingly.

In the second stage, an independent, blinded investigator will determine the presence of TLTV and LSTV, as well as the pathological disc level, using a sagittal whole-spine MRI localizer that includes the entire spinal axis from C2 to the sacrum. In the final analysis, the agreement between the two assessment methods will be examined. The study will determine the accuracy of level identification based on axial and sagittal lumbar MRI sequences and thoracolumbar/lumbosacral radiographs. Additionally, the detectability of lumbar ribs or rib agenesis based solely on radiographic findings will be evaluated. Finally, the true anatomical level corresponding to each marker will be identified using the whole-spine localizer and reported accordingly.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75 years
* Presenting to the outpatient clinic with low back and leg pain
* Diagnosis of lumbar radicular pain based on history, physical examination, and lumbar MRI findings
* Willingness and ability to provide informed consent to participate in the study

Exclusion Criteria:

* History of spinal surgery
* Patients with incomplete or unavailable medical records within the hospital information system

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will include adult patients aged 18 to 75 years who present to the outpatient Algology clinic with complaints of low back and leg pain. Participants must receive a clinical diagnosis of lumbar radicular pain based on history, physical examination, and lumbar MRI findings. Only patients with complete and accessible medical records will be included. Individuals with a history of spinal surgery will be excluded from the study.
  Sample size of the study: 250
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Accuracy of Vertebral Level Identification Using Routine Lumbar MRI | At the time of imaging evaluation (baseline)
  Accuracy of vertebral level identification based solely on routine lumbar MRI sequences (axial and sagittal), compared with whole-spine sagittal localizer imaging (gold standard). Accuracy will be calculated as the proportion of correctly identified pathological disc levels.
  How It Will Be Measured:
  Correct level matching (Yes/No) Accuracy (%) = (Correct identifications / Total cases) × 100

SECONDARY OUTCOMES:
Agreement Between MRI-Based Anatomical Landmarks and True Vertebral Levels | Baseline
  Agreement between each anatomical marker (aortic bifurcation, inferior vena cava bifurcation, right renal artery, conus medullaris) and the true vertebral level determined by whole-spine localizer imaging.
  Measurement: Cohen's kappa (κ), absolute level difference (levels above/below), mean ± SD
Frequency and Types of Transitional Vertebrae (LSTV and TLTV) | Baseline
  Prevalence and subtype distribution of lumbosacral transitional vertebrae (Castellvi classification) and thoracolumbar transitional vertebrae. Measurement: n (%) by subtype.
Effect of Transitional Vertebrae on Level Misidentification | Baseline
  Comparison of the misidentification rate of disc levels in patients with vs. without transitional vertebrae.
  Measurement: Misidentification rate (%), Relative risk, 95% CI

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara Üniversitesi Tıp Fakültesi, Istanbul, Maltepe, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No